CLINICAL TRIAL: NCT05404295
Title: The Effect of Treatment With Umbilical Cord Blood Platelet Lysate on Diabetic Foot Ulcers:a Randomized Controlled Trial
Brief Title: The Effect of Treatment With Umbilical Cord Blood Platelet Lysate on Diabetic Foot Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Attikon Hospital (Other)
Collaborators: Biomedical Research Foundation, Academy of Athens (Other)
Responsible Party: Principal Investigator, VAIA LAMBADIARI, Professor of Internal Medicine-Endocrinology, Attikon Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 411/05-06-2019
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical cord blood platelel lysate group (Active Comparator): A Umbilical cord blood platelel lysate gel will be applied in diabetic foot ulcer every three days for one month.
  Interventions: Other: Umbilical cord blood platelel lysate gel
- Control group (Placebo Comparator): The control group will receive the clinical standard of care; removable of any necrotic, hyperkeratotic and infected tissue, cleansing of the wound with normal saline and covering of the ulcer with dressing with normal saline and then with a few layers of sterile gauze, and non-compressible bandage.
  Interventions: Other: Umbilical cord blood platelel lysate gel

INTERVENTIONS:
Other: Umbilical cord blood platelel lysate gel — For the treatment group, a gel from Umbilical cord blood platelel lysat will be applied in the ulcer, and then a few layers of sterile gauze, and non-compressible bandage will be used to cover the wound/ulcer area.

SUMMARY:
Application of autologous Platelet Rich Plasma (PRP) has been a major breakthrough for the treatment of diabetic foot ulcers, as it provides the necessary growth factors which enhance tissue healing. Human umbilical cord blood platelet lysate (UCB-PL) contains a supraphysiological concentration of growth factors. The aim of the study is to evaluate the efficacy of umbilical cord blood platelet lysate (UCB-PL) gel for the treatment of diabetic foot ulcer.

DETAILED DESCRIPTION:
110 patients with diabetic foot ulcer will be randomized to receive UCB-PL gel or regular dressing with normal saline. The diabetic foot ulcers will be first debrided to remove any necrotic and infected tissues or hyperkeratotic skin. Afterward, the wound area will be cleaned thoroughly with normal saline. Ulcer length, width and surface will be measured before any study procedure. The UCB-PL gel in the treatment group and the dressing with normal saline in the control group will be applied in the ulcer, and then a few layers of sterile gauze, and non-compressible bandage will be used to cover the wound/ulcer area. This will be repeated every three days for one month. After the fist one month of treatment, the patients will be followed up for a period of 20 weeks post-treatment. Care and management efforts will be provided at each visit included cleansing and assessing of the wound, obtaining an interim wound history, including information regarding adverse events, concomitant medications and other aspects of care since the last visit. Ulcers will be photographed at two weeks, at four weeks, at two months, at four months and at six months.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years old
* patients with diabetic foot ulcer, foot ulcer located on the plantar, medial, or lateral aspect of the foot (including all toe surfaces)
* ulcer with area(length x width) measurement<30 cm2
* non-infected ulcers

Exclusion Criteria:

* pregnacy
* venous ulcers
* clinical signs and symptoms of infection
* exposure of bone, muscle, ligaments, or tendons and the presence of tunneling

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
The efficacy of UCB-PL in ulcer healing by assessing the change in ulcer size. | six months
  Primary endpoint was to investigate the efficacy of UCB-PL in ulcer healing by assessing the change in ulcer size over the six months follow-up by using the imito-measure application.

CONTACTS AND LOCATIONS:
Overall Officials: Vaia Lambadiari, Professor, Principal Investigator — General University Attikon Hospital
Locations (2):
- Greece (2):
  - Catherine Stavropoulos-Giokas, Athens, Attica
  - Vaia Lambadiari, Athens, Attica